CLINICAL TRIAL: NCT01651455
Title: Maintaining Lung Function in Cystic Fibrosis Patients: Evaluation and Comparison Between Two Decades in a Retrospective Monocentric Observational Study
Brief Title: Retrospective Observational Study to Compare Cystic Fibrosis Patients in Two Decades Before and After 2000
Acronym: MAESTRALE
Status: Completed | Type: Observational
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Collaborators: Medidata Solutions (Industry)
Responsible Party: Sponsor
Other Study IDs: MAESTRALE
Record Dates: First submitted 2012-07-25; First posted 2012-07-27 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Pseudomonas Aeruginosa
MeSH Terms: conditions — Cystic Fibrosis; Pseudomonas Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cohort first decade: Patients born between 01/01/1979 and 12/31/1984
- Cohort second decade: Patients born between 01/01/1991 and 12/31/1996

SUMMARY:
The purpose of this study is to describe two cohorts of cystic fibrosis patients treated in 2 different decades in terms of FEV1 (Forced Expiratory Volume in one second) maintenance.

DETAILED DESCRIPTION:
The purpose of this study is to describe two cohorts of cystic fibrosis patients treated in terms of FEV1 maintenance from the age of 10 to 15 before and after 2000.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Cystic Fibrosis diagnosed with neo-natal screening
* Patients born between 01/01/1979 and 12/31/1984 (Cohort 1)and patients born between 01/01/1991 and 12/31/1996 (Cohort 2)
* Patients with at least 2 FEV1 yearly measurements from the age of 10 to 15

Exclusion Criteria:

* Patients with malignant tumor
* Patients with meconium ileus
* Patients with transplantation (pneumectomy or lobectomy)
* Patients involved in any other clinical trial
* Patients moved to another Clinical Center

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients affected with Pseudomonas A. living in the N-E area of Italy.
Sampling Method: Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2012-09; Primary Completion 2013-03 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
To describe the difference in terms of FEV1 decline between two cohorts of cystic fibrosis patients | 5 years

SECONDARY OUTCOMES:
To identify clinical parameters or treatments correlated to FEV1 maintenance in two cohorts of cystic fibrosis patients | 5 years
To evaluate the number of patients with Pseudomonas Aeruginosa infection during observational period | 5 years
To describe length of time without Pseudomonas A. infection in non-colonized patients during observational period. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Baroukh Maurice Assael, Professor, Principal Investigator — U.O. Fibrosi Cistica Azienda Ospedaliera Verona
Locations (1):
- U.O. Azienda Ospedaliera, Verona, Veneto, Italy